CLINICAL TRIAL: NCT05133219
Title: The Effect of ıntensified Sensory-based Therapy on Upper Extremity Functions and Activities of Daily Living in Patients With Chronic Stroke
Brief Title: The Effect of ıntensified Sensory-based Therapy on Upper Extremity Functions and Activities of Daily Living
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Muhammed Rohat YAZICI, Researcher Assistant, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KOU-MRYAZİCİ-001
Record Dates: First submitted 2021-09-09; First posted 2021-11-24 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Stroke; Sensory Defect
MeSH Terms: conditions — Stroke | interventions — Occupational Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Research Group (Experimental): Participants will be received Intensified sensory therapy.
  Other: Occupational Therapy Activities of Daily Living Training
  Intervention: Other: Occupational therapy intervention
  Interventions: Other: Occupational Therapy
- Control Group (Experimental): Participants will be received Occupational Therapy.
  Other: Activities of Daily Living Training
  Interventions: Other: Occupational Therapy

INTERVENTIONS:
Other: Occupational Therapy — Occupational therapy is the only profession that helps people across the lifespan to do the things they want and need to do through the therapeutic use of daily activities (occupations). Occupational therapy practitioners enable people of all ages to live life to its fullest by helping them promote health, and prevent-or live better with-injury, illness, or disability.
  Other Names: Activities of Daily Living Training; İntensified Sensory Therapy

SUMMARY:
Sensory dysfunction following stroke is a common condition. The deficiency in the somatosensory system negatively affects the learning of new motor skills by preventing feedback from the sensory system, and it can also cause problems in daily life, personal care, productivity, and leisure activities. Somatosensory impairment is often overlooked, as rehabilitation often focuses on motor abilities in the affected extremity. In the studies reviewed, it is stated that sensory dysfunction is seen in approximately 50% of stroke patients.

The aim of this study is to examine the effects of intensified sensory-based therapy applied to the affected upper extremity sensory functions in individuals with chronic stroke on the upper extremity functions, quality of life, and independence of daily living activities.

DETAILED DESCRIPTION:
Sensory dysfunction following stroke is a common condition. The deficiency in the somatosensory system negatively affects the learning of new motor skills by preventing feedback from the sensory system, and it can also cause problems in daily life, personal care, productivity, and leisure activities. Somatosensory impairment is often overlooked, as rehabilitation often focuses on motor abilities in the affected extremity. In the studies reviewed, it is stated that sensory dysfunction is seen in approximately 50% of stroke patients.

The aim of the study; The aim of this study is to examine the effects of intensified sensory-based therapy applied to the affected upper extremity sensory functions in individuals with chronic stroke on the upper extremity functions, quality of life, and independence of daily living activities.

Thirty patients with chronic stroke will be randomized 1:1 to study (n:15) and control (n=12). Thumb localization test, finger swipe test, stereognosis test, and two-point discrimination test will be used to evaluate the sensory functions of individuals. Demographic information of individuals will be recorded with a sociodemographic information form. Before the treatment, the sensory levels of all patients will be determined by thumb localization, finger scrolling and stereognosy tests. Jebsen Taylor Hand Function Test (JTHFT), Modified Frenchay Scale (MFS), Canadian Occupational Performance Measure (COPM), Goal Attainment Scale (GAS) and Stroke-Specific Quality of Life Scale (SSQOL) will be administered before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Stroke duration more than 6 months,
* To be able to communicate
* 10 degrees of wrist dorsiflexion starting from full palmar flexion of the wrist
* To initiate finger extension

Exclusion Criteria:

* Joint contracture in the upper and lower extremities that will affect functionality other than stroke,
* Having a significant uncontrolled health problem and a history of epileptic seizures,
* Having 3 or more spasticity according to the Modified Ashworth Scale (MAS),
* Unable to communicate and cooperate,
* With marked ataxia and dystonia,
* Lack of movement and function in the wrist and fingers
* Having a diagnosis of bilateral stroke

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-05-23 (Actual); Primary Completion 2022-08-08 (Actual); Study Completion 2022-09-02 (Actual)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure (COPM)- Satisfaction | 3 weeks
  Used to evaluate participants' self-perceived satisfaction with performance. In this structured interview, participants are asked to select 5 tasks to perform and then rate their satisfaction of how well they are able to complete each task on a scale of 1 (unsatisfied) to 10 (completely satisfied). Total scores are an mean of individual task scores and also range from 1 (unsatisfied) to 5 (completely satisfied). Collected data will be used to measure changes within and between groups on self-perceived satisfaction with performance between week 1 and 8, week 1 and 3.
Canadian Occupational Performance Measure (COPM)- Performance | 3 weeks
  Used to evaluate participants' self-perceived functional performance. In this structured interview, participants are asked to select 5 tasks to perform and then rate their perception of how well they are able to complete each task on a scale of 1 (unable to perform) to 10 (able to perform extremely well). Total scores are an mean of individual task scores and also range from 1 (unable to perform tasks) to 5 (able to perform tasks extremely well). Collected data will be used to measure changes within and between groups on self-perceived performance between week 1 and 3.
Jebsen Taylor Hand Function Test (JTHFT) | 3 weeks
  The JTHFT is a common and detailed clinical assessment for fine motor skills with weighted and non-weighted hand functions. The test is derived from activities of daily routine and consists of writing a standardized sentence, turning over 5 cards, picking up and replacing small objects; simulated eating using a spoon and 5 kidney beans, stacking 4 draughts pieces on a board, turning over 5 large empty tins and turning over 5 full tins.
The Modified Frenchay Scale (MFS) | 3 weeks
  The Modified Frenchay Scale (MFS) measures active upper limb function in hemiparesis based on a video review of 10 everyday living tasks, each rated on a 10-point visual analogic scale. Six tasks are bimanual and four are unimanual performed with the paretic hand. We will measured intra- and inter-rater reliability of MFS in hemiparetic patients among trained raters.

SECONDARY OUTCOMES:
The Stroke Specific Quality Of Life Scale (SSQOL) | 3 weeks
  The Stroke Specific Quality Of Life scale (SS-QOL) is a patient-centered outcome measure intended to provide an assessment of health-related quality of life specific to patients with Stroke.
  To assess the quality of life of stroke patients, Williams et al. The Stroke Specific Quality of Life Scale (SSQOL) created by the Institute will be used. The SSQOL consists of 12 subsections, including energy, family roles, language, mobility, mood, personality, self-care, social roles, thinking, upper extremity function, vision and work/productivity, and a total of 49 questions; It is graded with a Likert-type scoring ranging from 1 to 5.
Sensory Test- Stereognosy Test | 3 weeks
  Patients can easily recognize when their eyes are closed; 12 objects including water bottle, glass, scissors, paper, key, pen, glove, ruler, telephone, ball, fork and spoon were evaluated according to their naming. Patients will be evaluated in 2 groups as normal recognizing 7-12 objects and decreased recognizing 7 or less objects.
Sensory Test- Finger Shift Test | 3 weeks
  By looking at the patient's ability to distinguish up and down passive movement of the proximal thumb joint while his eyes are closed; decreased and will be considered normal.
Sensory Test- Thumb Localization Test | 3 weeks
  The patient was asked to localize the affected side with his good hand while his eyes were closed; decreased and will be considered normal.
Goal Attainment Scaling (GAS) | 3 weeks
  GAS served as the primary outcome measure. Once a patient has identified a goal area, GAS goals are established using a 5-point scale, with ''0'' reflecting a score indicating the patient met his or her goal as expected; scores of +1 or +2 indicate surpassing the desired goal, and -1 or -2 indicate inadequate goal attainment. Each potential score (i.e. -2, -1, 0, +1, +2) is based on a criterion that is established collaboratively with the patient and is measurable and specific.

CONTACTS AND LOCATIONS:
Overall Officials: Çiğdem ÇEKMECE, PhD, Study Chair — Kocaeli University
Locations (1):
- Kocaeli Üniversitesi, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No